CLINICAL TRIAL: NCT05787184
Title: Sepsis Early Evaluation Through Rapid Ultrasound and Venous Gas Analysis: a Prospective Observational Study in the Emergency Department
Brief Title: Sepsis Early EvaluatioN Through Rapid Ultrasound and veNous Gas Analysis
Acronym: See'n'Run
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Fondazione Policlinico Universitario Agostino Gemelli IRCCS (Other)
Responsible Party: Principal Investigator, FRANCESCHI FRANCESCO, Professor Francesco Franceschi, Head of the Emergency Medicine Department, Fondazione Policlinico Universitario Agostino Gemelli IRCCS
Other Study IDs: 4925
Record Dates: First submitted 2023-02-27; First posted 2023-03-28 (Actual); Last update posted 2023-03-28 (Actual); Status verified 2023-03

CONDITIONS: Sepsis; Septic Shock; Shock
Keywords: ultrasound; echography; POCUS; venous blood gas; emergency medicine
MeSH Terms: conditions — Sepsis; Shock, Septic; Shock

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Sepsis is a life-threatening condition, caused by a systemic infection. It is particularly dangerous in already fragile populations and needs to be identified quickly to be treated as fast as possible, as discussed during the 2016 sepsis consensus and highlighted by the 2021 Surviving Sepsis Campaign. Yet, while there are scores to quickly identify patients who are at an increased risk of mortality (namely quick-SOFA, q-SOFA), these scores are also highly unspecific and cannot guarantee an adequate risk stratification. Therefore, it would be extremely valuable to further stratify mortality risk in patients who present to the emergency medical evaluation, especially those who present with stable hemodynamics but are at increased risk of decompensation during hospital stay. Furthermore, in the emergency room, it is sometimes impossible to re-evaluate patients regularly, thus, it would be important to immediately identify high-risk patients. Unfortunately, at the moment, there is no consensus. Through this study, the investigators will try to identify ultrasound parameters and biochemical markers which can be obtained during the first visit in the emergency room (ER) and that allow a quick risk stratification of patients with sepsis.

The rationale of this study is to improve early identification of septic patients who are at risk of rapid deterioration in the course of their permanence in the ER and the hospital wards in general. The investigators selected a number of clinical, laboratory and bedside ultrasound parameters which have been previously shown to be correlated with mortality in sepsis, and will seek to identify which among these parameters best correlates with prognosis when acquired in the very first minutes of a patient's arrival in the ER. The objective would be to analyse these parameters and eventually to propose a new early sepsis score which might help the emergency physician to better tailor its efforts and clinical resources to the most sick patients.

DETAILED DESCRIPTION:
The investigators propose a multicenter, prospective, observational study which will take place between January 2023 until the pre-specified target number of 400 patients is reached, in any case within 1 year, in three major urban, teaching Hospitals. At the end of the enrolling phase, data analysis and conclusion of the study will occur within 6 months.

These patients will undergo a regular emergency room (ER) visit, during which a venous blood gas and a bedside ultrasound will be obtained, along with the collection of anamnestic and clinical parameters. All of these procedures normally take place in the first medical evaluation in the ER, therefore no unnecessary procedures or harm to patients will take place.

The data which will be obtained during the first medical visit include:

Anamnestic and demographic data:

* Age;
* Sex;
* History of hypertension, diabetes, congestive heart failure, chronic lung disease, chronic kidney failure, severe immunosuppression, cancer;
* Infective source, if known or suspected.

Vital parameters:

* Glasgow Coma Scale (GCS) and AVPU scale;
* Systolic, diastolic and mean arterial blood pressure;
* Heart and respiratory rate;
* Body temperature;
* Capillary refill time (CRT);
* Peripheral oxygen saturation and oxygen supplementation if present.

Venous blood gas analysis:

* pH;
* glucose;
* lactate;
* hemoglobin;
* sodium and potassium.

Bedside ultrasound examination:

* inferior vena cava distensibility through visual gestalt;
* global left ventricular contractility through visual gestalt;
* mitral annular plane systolic excursion (MAPSE), obtained through apical 4-chamber view.

All the above mentioned data will be obtained and reported in a specific module and subsequently added to the database.

Following the first medical visit, patients will prosecute their clinical course with diagnostic and therapeutic strategies as chosen by the attending emergency physicians. No additional maneuvers will take place as far as study procedures are concerned.

After a week from the enrollment, two physicians responsible for the study procedures (L.F. and G.T.) will manually extract clinical and laboratory data concerning the enrolled patients from the digital Health System softwares of the involved Hospitals. Data concerning death during hospital stay, ICU or regular ward admission, laboratory values, eventual positivity of blood culture, etc will be obtained and added to the study database.

The data which will be obtained at a week from enrollment are:

* Patient outcome: mortality, ICU or general ward admission;
* Results of blood cultures or other cultures from relevant specimens, if available;
* Results of blood tests performed during the first evaluation in the ER, including: white blood cell count (WBC), hematocrit, creatinine, C-reactive protein (CRP), Procalcitonin.

The last set of data concerning mortality will be obtained at 30 days, whether in-hospital (through the electronic hospital record) or out-of-hospital by telephone call.

ELIGIBILITY:
Inclusion Criteria:

* All adult, non pregnant patients admitted to the ED with a clinical suspicion of sepsis or septic shock

Exclusion Criteria:

* Age less than 18 years old
* Pregnancy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: All patients who are admitted to the ED with a clinical suspicion of sepsis and septic shock at the first medical visit.
Sampling Method: Probability Sample
Enrollment: 400 (Estimated)
Dates: Start 2023-01-01 (Actual); Primary Completion 2024-01-01 (Estimated); Study Completion 2024-06-01 (Estimated)

PRIMARY OUTCOMES:
Number of participants who are dead for any cause | 7 days
  categorical variable

SECONDARY OUTCOMES:
Number of participants who die during the emergency department visit | 48 hours
  categorical variable
Number of participants who are dead for any cause | 30 days
  categorical variable
Number of patients who require ICU admission | 30 days
  categorical variable
Length of hospitalisation | 6 months
  continuous variable

CONTACTS AND LOCATIONS:
Locations (1):
- Fondazione Policlinico Universitario "A. Gemelli", IRCCS; Emergency Department, Rome, Lazio, Italy

IPD SHARING:
Plan to Share IPD: No